CLINICAL TRIAL: NCT06928116
Title: Physical Rehabilitation of Long COVID by Heat Therapy
Brief Title: Heat thErapy And mobiLity in COVID-19 Survivors
Acronym: HEAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0550-24-FB; R01AG089307 (NIH)
Record Dates: First submitted 2025-04-09; First posted 2025-04-15 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-07

CONDITIONS: Long COVID
Keywords: Heat Therapy; mobility limitations; Post-acute sequelae of SARS-CoV-2 infection (PASC)
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Hyperthermia; Mobility Limitation | interventions — Diathermy; Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Heat Therapy (Experimental): At home heat therapy 5 times (40-55 min) per week for 8 weeks.
  Interventions: Behavioral: Heat therapy
- Control Therapy (Sham Comparator): Sham at home thermoneutral therapy 5 times (40-55 min) per week for 8 weeks.
  Interventions: Behavioral: Sham Control
- Walking Intervention Using Wearable Technology (Active Comparator): +1,500-3000 steps per day 3-5 days a week for 8 weeks.
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Heat therapy — At home lower body heat therapy
  Arms: Heat Therapy
Behavioral: Sham Control — Sham Thermoneutral
  Arms: Control Therapy
Behavioral: Walking — Walking intervention
  Arms: Walking Intervention Using Wearable Technology

SUMMARY:
Post-acute sequelae of SARS-CoV-2 infection (PASC) is becoming a major risk factor for chronic diseases, with older adults and those with underlying health conditions at risk of developing persistent mobility limitations and disabilities. Although exercise intervention is a common strategy to restore functional capacity, it may not be feasible or enticing to many people with PASC. This clinical trial seeks to establish the tolerability and efficacy of at home lower-body heat therapy for improving functional capacity along with metabolic and vascular health in late-middle aged and older adults with PASC, also known as "long COVID".

DETAILED DESCRIPTION:
Post-acute sequelae of SARS-CoV-2 infection (PASC) affects 5 out of 10 patients hospitalized for the coronavirus disease 2019 (COVID-19) and ~11% of all adults infected by SARS-CoV-2, which makes this condition a growing public health concern. It is associated with important disabilities, cognitive dysfunction, and increased risks for cardiovascular and metabolic diseases. Although exercise-based intervention is a promising rehabilitation strategy, participation rates are commonly low in clinical population. In addition, post-exertional malaise, a common symptom with PASC, is a major safety concern in these patients, which may prevent a significant proportion of these individuals to receive adequate rehabilitation. In this context, there is a critical need to develop well-tolerated and effective strategies at home that ameliorates health and functional capacity in individuals with PASC. One promising approach that offers numerous health benefits is whole-body heat therapy. Whether this intervention is effective when confined to the lower body and well tolerated at home in people with PASC is, however, unknown.

The overall objective of this project is to determine the safety, tolerability, and efficacy of home-based lower body heat therapy in late middle-age and older adults with PASC. Investigators will test the central hypothesis that home-based lower body heat therapy is safe, well adhered, and can improve functional capacity and several surrogate markers for metabolic and vascular health in late-middle age and older adults with PASC. Specific Aim 1 will test the hypothesis that lower body heat therapy at home is safe, well adhered, and improve both cognitive and physical function in middle-age and older adults with PASC. Selected participants will be randomly allocated to perform 8 weeks of home-based lower body heat therapy (HT, skin temperature 38-40˚C, 40-55 min, 5 per week at home), a thermoneutral condition (CT, skin temperature 33˚C, same duration and frequency), or a walking intervention using wearable technology (WT, 1,500-3,000 additional steps from baseline, 3-5 days per week). We will compare the 6 min walking distance, the short physical performance battery test score, gait speed, cognitive function, incidence of adverse events, and participant's adherence to intervention between groups. Specific Aim 2 will test the hypothesis that heat therapy will attenuate inflammation, which will then decrease arterial stiffness, and improve both vascular endothelial function and muscle intracellular oxygen availability in participants with PASC. Investigators will use in vitro assays on blood samples and Doppler ultrasound techniques to assess changes in inflammation, redox status, pulse-wave velocity, and flow-mediated dilation. Muscle intracellular oxygen availability will be measured by magnetic resonance spectroscopy in vivo. Specific Aim 3 will test the hypothesis that lower body heat therapy will improve glucose control as a result of enhanced mitochondrial function. All these effects will not be statistically inferior to the WT group. The proposed research is highly significant as it is easily translatable and is expected to guide future rehabilitation strategies to mitigate long-term disabilities in patients with PASC.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 50 and 90 years
* Free from orthopedic limitations that would prohibit performing leg exercise
* BMI < 40 kg/m2 and weigh < 400lbs
* Previously contracted Covid-19 and have persistent symptoms such as a fatigue or decline in physical function, for at least 2 months following SARS-CoV-2 infection

Exclusion Criteria:

* Unable to give written informed consent
* Women who are pregnant, breastfeeding, or likely to become pregnant within the next 6 months
* Women who are taking hormone therapy
* Claustrophobia
* Orthopedic limitations that would prohibit them from walking
* Currently enrolled in an exercise-based or respiratory muscle rehabilitation program.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
6 min walking distance | 8 weeks
  Distance covered during 6 min of walking
Short Physical Performance Battery Test | 8 weeks
  Test of physical functional capacity
Arterial stiffness | 8 weeks
  Pulse Wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Gwenael Layec, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data will be deposited into a Data Repository specific to biomedical sciences using standard rights waivers as those established by Open Data Commons (ODC)
Supporting Information: Study Protocol
Time Frame: The research community will have access to data at the end of the grant award or when a publication has been submitted, whichever comes first.
Access Criteria: Data will be deposited on open access platform and we will use standard rights waivers established by Open Data Commons (ODC).